CLINICAL TRIAL: NCT05070494
Title: Efficacy of Different Doses of Influenza Vaccine in Chronic Hemodialysis Patients: Randomized Controlled Trial (Enhance Study)
Brief Title: Efficacy of Different Doses of Influenza Vaccine in Chronic Hemodialysis Patients
Acronym: Enhance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Bhumirajanagarindra Kidney Institute, Thailand (Other); Ministry of Health, Thailand (Other Government)
Responsible Party: Principal Investigator, Angsana Phuphuakrat, Angsana Phuphuakrat, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MURA2019/1116
Record Dates: First submitted 2021-09-04; First posted 2021-10-07 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: ESRD; Influenza Vaccine; Seroprotection
Keywords: ESRD; Influenza vaccine; double dose Influenza vaccine; double dose booster Influenza vaccine; Immune response
MeSH Terms: conditions — Kidney Failure, Chronic; Influenza, Human | interventions — Influenza Vaccines; Antigens, Surface

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ้healthy subject with standard dose trivalent influenza vaccine (Other): ้healthy volunteer that received Egg-derived standard dose trivalent influenza vaccine (surface antigen, inactivated) ( 0.5 ml : 15 mcg/strain)
  Interventions: Biological: Egg-derived standard dose trivalent influenza vaccine (surface antigen, inactivated)
- ESRD patient with standard dose trivalent influenza vaccine (Active Comparator): ESRD patient that received Egg-derived standard dose trivalent influenza vaccine (surface antigen, inactivated) ( 0.5 ml : 15 mcg/strain)
  Interventions: Biological: Egg-derived standard dose trivalent influenza vaccine (surface antigen, inactivated)
- ESRD patient with double dose trivalent influenza vaccine (Experimental): ESRD patient that received Egg-derived double dose trivalent influenza vaccine (surface antigen, inactivated) total 1 ml ( 1 ml /(30 mcg/strain)
  Interventions: Biological: Egg-derived standard dose trivalent influenza vaccine (surface antigen, inactivated)
- ESRD patient with double dose - booster trivalent influenza vaccine (Experimental): ESRD patient that received Egg-derived double dose trivalent influenza vaccine (surface antigen, inactivated) ( 1 ml /(30 mcg/strain) and booster with Egg-derived double dose trivalent influenza vaccine (surface antigen, inactivated) ( 1 ml /(30 mcg/strain) at next 6 months after first dose
  Interventions: Biological: Egg-derived standard dose trivalent influenza vaccine (surface antigen, inactivated)

INTERVENTIONS:
Biological: Egg-derived standard dose trivalent influenza vaccine (surface antigen, inactivated) — study of immunologic response to different dose and duration of Egg-derived standard dose trivalent influenza vaccine (surface antigen, inactivated)

SUMMARY:
This study was a randomized controlled trial to investigate the immune response of influenza vaccines when doses were increased. and a second vaccination together with an increase in the amount of vaccine in patients with chronic kidney disease receiving hemodialysis

DETAILED DESCRIPTION:
1. Patients with chronic kidney disease undergoing dialysis will be examined by an internist.
2. Collect the necessary basic information of patients who agree to participate in the treatment.
3. Patients will be randomized to be divided into 3 groups: those who will receive an standard dose of influenza vaccine, those who will receive double standard dose of influenza vaccine (double-dose) and those who will receive double standard dose of influenza vaccine and Six months after the first dose of vaccination (double-booster-dose), 50 people per group.
4. Non-dialysis volunteers will be invited to participate in the research. to be a control group of 25 people
5. Patients with chronic kidney disease and volunteers will receive basic laboratory blood tests.
6. Patients with chronic kidney disease and volunteers will be vaccinated against influenza. shoulder muscle area according to random groups The details of using Influvac vaccine of that year are produced by Abbott.
7. Patients with chronic kidney disease and volunteers are asked about the potential side effects of vaccination. according to research guidelines both systemic side effects and injection site Each time receiving hemodialysis 3 times a week for 2 weeks after vaccination
8. Patients with chronic kidney disease and volunteers were asked about the onset of symptoms of respiratory infection throughout the 12-month study period after vaccination.
9. Patients will receive a blood test to check their immune response to influenza vaccine. (Hemagglutination inhibition assays and activation and/or exhaustion T cell markers, T cell subpopulation by flow cytometry) at 1, 6, 7 and 12 months after influenza vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Received kidney replacement therapy with dialysis for more than 1 month.
* Hemodialysis at least 3 times a week
* (Kt/v) greater than 1.2
* Never received an organ transplant.
* Life expectancy of more than 1 year
* Research participants or representatives are welcome to join the project by signing.

Exclusion Criteria:

* History of any vaccinations in the 4 weeks prior to the study.
* History of receiving influenza vaccine 6 months before entering this study.
* History of allergy to flu vaccine or allergic to egg white
* Fever or headache, muscle pain (influenza-like illness) 3 days before vaccination
* Thrombocytopenia
* On immunosuppressive drug (Prednisolone 15 mg daily or equivalent for two weeks in a row in the previous 3 months) or immunocompromised patient
* Patient or family history of having had Guillain-Barre disease. (Guillain-Barre syndrome)
* The research participant or his representative refuses or requests to withdraw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
To compare proportion of seroprotection of different doses of influenza vaccine in hemodialysis patients at month 12 | 12 months
  Patients will receive a blood test to check their immune response to influenza vaccine. (Hemagglutination inhibition assays and activation and/or exhaustion T cell markers, T cell subpopulation by flow cytometry) at month 12 after influenza vaccination.

SECONDARY OUTCOMES:
To compare the prevention of influenza virus infection in different doses of influenza vaccination. | 12 months of data collection
  to compare incidence rate of influenza infection in different doses of influenza

CONTACTS AND LOCATIONS:
Locations (1):
- Angsana Phuphuakrat, Ratchathewi, ฺBangkok, Thailand

REFERENCES:
- [Background] Chou CY, Wang SM, Liang CC, Chang CT, Liu JH, Wang IK, Hsiao LC, Muo CH, Huang CC, Wang RY. Risk of pneumonia among patients with chronic kidney disease in outpatient and inpatient settings: a nationwide population-based study. Medicine (Baltimore). 2014 Dec;93(27):e174. doi: 10.1097/MD.0000000000000174. PMID 25501062
- [Background] Collins AJ, Foley RN, Gilbertson DT, Chen SC. The state of chronic kidney disease, ESRD, and morbidity and mortality in the first year of dialysis. Clin J Am Soc Nephrol. 2009 Dec;4 Suppl 1:S5-11. doi: 10.2215/CJN.05980809. PMID 19996006
- [Background] Viasus D, Garcia-Vidal C, Cruzado JM, Adamuz J, Verdaguer R, Manresa F, Dorca J, Gudiol F, Carratala J. Epidemiology, clinical features and outcomes of pneumonia in patients with chronic kidney disease. Nephrol Dial Transplant. 2011 Sep;26(9):2899-906. doi: 10.1093/ndt/gfq798. Epub 2011 Jan 27. PMID 21273232
- [Background] Sarnak MJ, Jaber BL. Pulmonary infectious mortality among patients with end-stage renal disease. Chest. 2001 Dec;120(6):1883-7. doi: 10.1378/chest.120.6.1883. PMID 11742917
- [Background] Cohen G, Horl WH. Immune dysfunction in uremia—an update. Toxins (Basel). 2012 Oct 24;4(11):962-90. doi: 10.3390/toxins4110962. PMID 23202302
- [Background] Girndt M, Sester M, Sester U, Kaul H, Kohler H. Molecular aspects of T- and B-cell function in uremia. Kidney Int Suppl. 2001 Feb;78:S206-11. doi: 10.1046/j.1523-1755.2001.59780206.x. PMID 11169012
- [Background] Anding K, Gross P, Rost JM, Allgaier D, Jacobs E. The influence of uraemia and haemodialysis on neutrophil phagocytosis and antimicrobial killing. Nephrol Dial Transplant. 2003 Oct;18(10):2067-73. doi: 10.1093/ndt/gfg330. PMID 13679482
- [Background] Lim WH, Kireta S, Leedham E, Russ GR, Coates PT. Uremia impairs monocyte and monocyte-derived dendritic cell function in hemodialysis patients. Kidney Int. 2007 Nov;72(9):1138-48. doi: 10.1038/sj.ki.5002425. Epub 2007 Aug 29. PMID 17728708
- [Background] Sester U, Sester M, Hauk M, Kaul H, Kohler H, Girndt M. T-cell activation follows Th1 rather than Th2 pattern in haemodialysis patients. Nephrol Dial Transplant. 2000 Aug;15(8):1217-23. doi: 10.1093/ndt/15.8.1217. PMID 10910448
- [Background] Fernandez-Fresnedo G, Ramos MA, Gonzalez-Pardo MC, de Francisco AL, Lopez-Hoyos M, Arias M. B lymphopenia in uremia is related to an accelerated in vitro apoptosis and dysregulation of Bcl-2. Nephrol Dial Transplant. 2000 Apr;15(4):502-10. doi: 10.1093/ndt/15.4.502. PMID 10727545
- [Background] Meier P, Golshayan D, Blanc E, Pascual M, Burnier M. Oxidized LDL modulates apoptosis of regulatory T cells in patients with ESRD. J Am Soc Nephrol. 2009 Jun;20(6):1368-84. doi: 10.1681/ASN.2008070734. Epub 2009 Apr 30. PMID 19406979 (Retraction: PMID 24459234 J Am Soc Nephrol. 2014 Mar;25(3):645)
- [Background] Wang IK, Lin CL, Lin PC, Liang CC, Liu YL, Chang CT, Yen TH, Morisky DE, Huang CC, Sung FC. Effectiveness of influenza vaccination in patients with end-stage renal disease receiving hemodialysis: a population-based study. PLoS One. 2013;8(3):e58317. doi: 10.1371/journal.pone.0058317. Epub 2013 Mar 13. PMID 23516462
- [Background] McGrath LJ, Kshirsagar AV, Cole SR, Wang L, Weber DJ, Sturmer T, Brookhart MA. Influenza vaccine effectiveness in patients on hemodialysis: an analysis of a natural experiment. Arch Intern Med. 2012 Apr 9;172(7):548-54. doi: 10.1001/archinternmed.2011.2238. PMID 22493462
- [Background] Gilbertson DT, Unruh M, McBean AM, Kausz AT, Snyder JJ, Collins AJ. Influenza vaccine delivery and effectiveness in end-stage renal disease. Kidney Int. 2003 Feb;63(2):738-43. doi: 10.1046/j.1523-1755.2003.00787.x. PMID 12631142
- [Background] Grohskopf LA, Sokolow LZ, Olsen SJ, Bresee JS, Broder KR, Karron RA. Prevention and Control of Influenza with Vaccines: Recommendations of the Advisory Committee on Immunization Practices, United States, 2015-16 Influenza Season. MMWR Morb Mortal Wkly Rep. 2015 Aug 7;64(30):818-25. doi: 10.15585/mmwr.mm6430a3. PMID 26247435
- [Background] Centers for Disease Control and Prevention (CDC). Prevention and control of seasonal influenza with vaccines. Recommendations of the Advisory Committee on Immunization Practices--United States, 2013-2014. MMWR Recomm Rep. 2013 Sep 20;62(RR-07):1-43. PMID 24048214
- [Background] Rubin LG, Levin MJ, Ljungman P, Davies EG, Avery R, Tomblyn M, Bousvaros A, Dhanireddy S, Sung L, Keyserling H, Kang I; Infectious Diseases Society of America. 2013 IDSA clinical practice guideline for vaccination of the immunocompromised host. Clin Infect Dis. 2014 Feb;58(3):309-18. doi: 10.1093/cid/cit816. PMID 24421306
- [Background] DiazGranados CA, Dunning AJ, Robertson CA, Talbot HK, Landolfi V, Greenberg DP. Efficacy and immunogenicity of high-dose influenza vaccine in older adults by age, comorbidities, and frailty. Vaccine. 2015 Aug 26;33(36):4565-71. doi: 10.1016/j.vaccine.2015.07.003. Epub 2015 Jul 14. PMID 26187260
- [Background] Rautenberg P, Proppe D, Schutte A, Ullmann U. Influenza subtype-specific immunoglobulin A and G responses after booster versus one double-dose vaccination in hemodialysis patients. Eur J Clin Microbiol Infect Dis. 1989 Oct;8(10):897-900. doi: 10.1007/BF01963779. PMID 2512137
- [Background] Liao Z, Xu X, Liang Y, Xiong Y, Chen R, Ni J. Effect of a booster dose of influenza vaccine in patients with hemodialysis, peritoneal dialysis and renal transplant recipients: A systematic literature review and meta-analysis. Hum Vaccin Immunother. 2016 Nov;12(11):2909-2915. doi: 10.1080/21645515.2016.1201623. Epub 2016 Jul 8. PMID 27392026
- See also: Related Info — https://immunityageing.biomedcentral.com/articles/10.1186/1742-4933-9-19
- See also: Related Info — https://www.cdc.gov/mmwr/preview/mmwrhtml/mm5916a2.htm